CLINICAL TRIAL: NCT01485588
Title: A Phase 1 / 2 Trial to Investigate The Safety and Tolerability of Single and Repeated Doses of hI-CON1™ Following Administration by Intravitreal Injection in Subjects With Neovascular Age-Related Macular Degeneration (AMD)
Brief Title: Safety and Tolerability Study for Age-Related Macular Degeneration
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Iconic Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IT-001
Record Dates: First submitted 2011-12-01; First posted 2011-12-05 (Estimated); Results first posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-10

CONDITIONS: Neovascular Age-Related Macular Degeneration
MeSH Terms: interventions — hI-con1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- hI-con1™ 60µl (Experimental): Phase 1- This is a dose escalation study (60µl, 150µl, or 300 µl) given at baseline and then the subject is followed up to week 24.
  Interventions: Drug: hI-con1™ 60µl
- hI-con1™ 150µl (Experimental): Phase 1- This is a dose escalation study (60µl, 150µl, or 300 µl) given at baseline and then the subject is followed up to week 24.
  Interventions: Drug: hI-con1™ 150µl
- hI-con1™ 300µl (Experimental): Phase 1- This is a dose escalation study (60µl, 150µl, or 300 µl) given at baseline and then the subject is followed up to week 24.
  Interventions: Drug: hI-con1™ 300µl

INTERVENTIONS:
Drug: hI-con1™ 60µl — Phase 1: 60µl, 150µl, or 300µl per injection (in the eye) on Day 1 only
  Arms: hI-con1™ 60µl
Drug: hI-con1™ 150µl — Phase 1: 60µl, 150µl, or 300µl per injection (in the eye) on Day 1 only
  Arms: hI-con1™ 150µl
Drug: hI-con1™ 300µl — Phase 1: 60µl, 150µl, or 300µl per injection (in the eye) on Day 1 only
  Arms: hI-con1™ 300µl

SUMMARY:
Phase 1: The purpose of this study is to evaluate the safety and tolerability of single ascending doses of hI-con1™ for subjects with Age-Related Macular Degeneration.

Phase 2: The purpose of this study is to evaluate the safety of 3 injections of hI-con1™ at 2 different dose levels.

ELIGIBILITY:
Ocular Inclusion Criteria:

* Active choroidal neovascularization (CNV) associated with age-related macular degeneration, as evidenced on fluorescein angiography (FA) and Optical Coherence Tomography (OCT), with the following lesion characteristics:
* Subretinal hemorrhage if present < 50% of total lesion size
* During Phase 1, the 4th, 5th, and 6th subjects enrolled in each cohort must have total lesion area < 6 Disc Area (DA) (total area of detachment) (15.24 mm2), of which at least 50% must be actively leaking, and 30% should be classic on the angiography as determined by a reading center, and no more than 3 prior injections of any therapy for the treatment of CNV.
* For Phase 2, total lesion area < 6 DA (total area of detachment) (15.24 mm2), of which at least 50% must be actively leaking, and 30% should be classic on the angiography as determined by a reading center and no more than 3 prior injections of any therapy for the treatment of CNV.
* Best Corrected Visual Acuity (BCVA) for Phase 1: 20/ 80 - count fingers in the study eye; visual acuity in the fellow eye must be the same or better than the study eye
* BCVA for Phase 2: 20/40 to 20/320 in the study eye; visual acuity in the fellow eye must be the same or better than the study eye
* Only one eye of each subject will be treated in the study. If both eyes are eligible, the study eye will be the eye with the worst visual acuity. If visual acuity is the same in both eyes, the eye with the most active CNV will be selected to be the study eye
* Clear ocular media and adequate pupillary dilation in the study eye to permit fundus photography for screening
* Intraocular pressure of 21 mm Hg or less in the study eye.

General Inclusion Criteria

* Subjects of either gender, > 50 years of age
* Subjects who are informed of, and willing and able to comply with, the investigational nature of the study and are able to provide written informed consent
* Ability to return for all study visits
* Females must be of non-child bearing potential (surgically sterilized or at least 2 years post-menopausal) or if of child-bearing potential, the subject must have a negative serum pregnancy test within 14 days prior to the first injection and agree to use 2 forms of effective contraception during the trial and for at least 60 days following the last study injection.

Ocular Exclusion Criteria:

* Any retinal vascular disease or retinal degeneration other than AMD in the study eye
* Serous pigment epithelial detachment without the presence of choroidal neovascularization in the study eye
* Pigment epithelial tears or rips in the study eye
* Previous posterior vitrectomy or retinal surgery in the study eye
* Any periocular infection in the past 4 weeks in the study eye
* During the duration of the study, subjects cannot be on any concomitant therapy with anti-VEGF (Vascular Endothelial Growth Factor) agents, e.g., Lucentis® , Avastin®, or Macugen® in the study eye (unless identified as rescue therapy given according to protocol guidelines)
* Concomitant therapy or use within 30 days of Baseline (Day 1) of systemic (e.g. intravenous, oral, intramuscular, rectal) corticosteroids in doses > 10 mg/ day prednisone or prednisone equivalent, or use of intravitreous or periocular steroids within 90 days of Baseline (Day 1) in the study eye
* Any current or prior use of extended-release steroid implants (e.g., Retisert®, Posurdex®, Medidur®) in the study eye
* Significant media opacities, including cataract, in the study eye which might interfere with visual acuity, assessment of toxicity, or fundus photography.
* Cataract surgery in the study eye within three months of screening
* Trabeculectomy or outflow-device glaucoma surgery in the study eye
* Intraocular surgery in the study eye within three months of screening
* Periocular or ocular infection in the study eye
* Severe myopia (spherical equivalent -8 diopters or greater) in the study eye
* History of vascular pigment epithelial detachment or submacular hemorrhage in the fellow eye.

General Exclusion Criteria:

* Use of any investigational agent or participation in any clinical trial of an investigational agent or investigational therapy that has the potential to affect the disease process (neovascular AMD) in the study eye within sixty (60) days of Baseline (Day 1), or participation in any other clinical trial of an investigational agent or investigational therapy within thirty (30) days of Baseline (Day 1). Participation in clinical trials of oral supplements of vitamins and minerals for the prevention of neovascular AMD (e.g. AREDS2) are allowed, as are studies that do not involve the administration of an investigational agent and/or investigational therapy
* Undiagnosed acute illness first observed during screening or between screening and baseline, or severe concurrent medical conditions that, in the investigator's judgment, represent a safety concern.
* Allergy to or prior significant adverse reaction to fluorescein
* Any major surgical procedure within one month of trial entry
* Blood pressure >160/90 mmHg.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-12; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Rocky Mountain Eye Center, P.C., Missoula, Montana
  - Retina & Vitreous Center of Southern Oregon, P.C., Ashland, Oregon
  - Palmetto Retina Center, West Columbia, South Carolina
  - Retina Research Center, Austin, Texas
  - Valley Retina Institute, PA, McAllen, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- hI-con1™ 60µg; hI-con1™ 150µg; hI-con1™ 300µg: Phase 1- This is a dose escalation study 60µg, 150µg, or 300 µg) given at baseline and then the subject is followed up to week 24.
  hI-con1™: Phase 1: 60µg, 150µg, or 300µg per injection (in the eye) on Day 1 only
Period: Overall Study
Arm/Group | hI-con1™ 60µg | hI-con1™ 150µg | hI-con1™ 300µg
Started | 6 | 6 | 6
Completed | 6 | 6 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- hI-con1™ 60µg; hI-con1™ 150µg; hI-con1™ 300µg: This is a dose escalation study 60µg, 150µg, or 300 µg) given at baseline and then the subject is followed up to week 24.
- Total: Total of all reporting groups
Arm/Group | hI-con1™ 60µg | hI-con1™ 150µg | hI-con1™ 300µg | Total
Number analyzed (Participants) | 6 | 6 | 6 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 6 | 6 | 6 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4 | 8
  Male | 5 | 3 | 2 | 10
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Central Retinal Subfield Thickness as Measured by Optical Coherence Tomography (OCT) at Week 24 From Baseline
Description: The Mean Change in Central Retinal Subfield Thickness as Measured by OCT is part of the evaluation on the safety and tolerability of single ascending doses of hI-con1 and to assist in determining the Maximum Tolerated Dose (MTD) that can be administered by intravitreal injection.
Time Frame: 24 Weeks
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | hI-con1™ 60µg | hI-con1™ 150µg | hI-con1™ 300µg
Number analyzed (Participants) | 6 | 6 | 6
Microns | -98 (141.19) | -66 (42.03) | -180.8 (97.9)

2. Primary Outcome: Mean Change in Best Corrected Visual Acuity (BCVA) at Week 24 From Baseline
Description: The Mean Change in Best Corrected Visual Acuity (BCVA) is part of the evaluation on the safety and tolerability of single ascending doses of hI-con1 and to assist in determining the Maximum Tolerated Dose (MTD) that can be administered by intravitreal injection. BCVA is measured using the Early Diabetic Retinopathy Study (EDTRS) chart. More letters read result in a higher score.
Time Frame: 24 Weeks
Measure: Mean (Standard Deviation); unit: Letters
Groups:
- hI-con1™ 20µg; hI-con1™ 150µg; hI-con1™ 300µl: Phase 1- This is a dose escalation study 60µg, 150µg, or 300 µg) given at baseline and then the subject is followed up to week 24.
  hI-con1™: Phase 1: 60µg, 150µg, or 300µg per injection (in the eye) on Day 1 only
Arm/Group | hI-con1™ 20µg | hI-con1™ 150µg | hI-con1™ 300µl
Number analyzed (Participants) | 6 | 6 | 6
Letters | -9.3 (6.81) | 6.0 (1.00) | 15.7 (5.03)

ADVERSE EVENTS:
Arm/Group | hI-con1™ 60µg | hI-con1™ 150µg | hI-con1™ 300µg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 1/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | hI-con1™ 60µg (N=6) | hI-con1™ 150µg (N=6) | hI-con1™ 300µg (N=6)
Premature Atrial Contractions (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | hI-con1™ 60µg (N=6) | hI-con1™ 150µg (N=6) | hI-con1™ 300µg (N=6)
Anterior Chamber Cell (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctival Haemorrhage (Eye disorders) | 1 (1) | 2 (2) | 2 (2)
ConjunctivalHyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctival Oedema (Eye disorders) | 0 (0) | 2 (2) | 1 (1)
Corneal Epithelium Defect (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Detachment of Retinal Pigment Epithelium (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Eye Irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye Pain (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Eye Pruritus (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Macular Degeneration (Eye disorders) | 0 (0) | 1 (1) | 2 (2)
Retinal Dystrophy (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal Exudates (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal Haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Retinal Pigment Epithelial Tear (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Subretinal Fibrosis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vision Blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Visual Acuity Reduced (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vitreous Floaters (Eye disorders) | 0 (0) | 1 (1) | 2 (3)
Vitritis (Eye disorders) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No